CLINICAL TRIAL: NCT04646226
Title: A Randomized Trial of Fistula vs. Graft Arteriovenous Vascular Access in Older Adults With End-Stage Kidney Disease on Hemodialysis
Brief Title: The Arteriovenous Vascular (AV) ACCESS Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00069593; 1R01AG071803-01 (NIH)
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: End-Stage Kidney Disease; Hemodialysis Complication
Keywords: Hemodialysis; End-Stage Kidney Disease; central venous catheters; arteriovenous fistula [AVF]; arteriovenous graft [AVG]; Arteriovenous Vascular Access
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Study will determine if placement of a graft access will be more effective at having access switched from catheter to using the graft; have fewer interventions on the graft access; have better arm function; have better self-sufficiency with daily activities; and better quality of life compared to those who receive a fistula - identify strategies that decrease dialysis access failure and improve quality of life
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- fistula surgically placed (Experimental): Randomized group to have surgically placed fistula for permanent hemodialysis access
  Interventions: Procedure: surgical intervention for creation of a fistula
- graft surgically placed (Active Comparator): Randomized group to have surgically placed graft for permanent hemodialysis access
  Interventions: Device: AV graft

INTERVENTIONS:
Device: AV graft — The purpose of the surgery is to connect a large vein in the arm to a nearby artery indirectly by inserting a graft material (graft surgery)
  Arms: graft surgically placed
Procedure: surgical intervention for creation of a fistula — The purpose of the surgery is to connect a large vein in the arm to a nearby artery directly (fistula surgery)
  Arms: fistula surgically placed

SUMMARY:
This study is to prospectively compare the effectiveness and safety of the two types of arteriovenous access placement (fistula or graft) in older adults with end stage kidney disease and multiple chronic conditions

DETAILED DESCRIPTION:
This study will determine the effects of arteriovenous (AV) fistula versus AV graft vascular access strategy on the rate of catheter-free dialysis days and access-related infections - costs associated with the dialysis vascular access - patient-reported satisfaction with different processes of vascular access care (catheter, fistula, or graft) - and the relationship between preoperative functional status and incidence of fistula or graft maturation failure

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* End-stage kidney disease on hemodialysis via a central venous catheter
* Hemodialysis is the long-term modality of treatment for end-stage kidney disease
* Central venous catheter is the sole vascular access used for hemodialysis at the time of referral for arteriovenous access creation
* Referred by patient's nephrologist for placement of arteriovenous access
* At least one of the following comorbid conditions: cardiovascular disease, peripheral vascular disease, and/or diabetes mellitus
* Medically and surgically eligible to undergo surgical placement of an arteriovenous access, deemed by the treating healthcare providers
* Native vasculature deemed preoperatively to be suitable for surgical creation of either type of arteriovenous access (arteriovenous fistula or arteriovenous graft) in the opinion of the surgeon
* Patient agreed to study participation and signed the informed consent

Exclusion Criteria:

* Severe cardiac disease defined as presence of either of the following three conditions: congestive heart failure with ejection fraction ≤ 20%, heart transplant, or ventricular assist device
* Known or suspected central vein stenosis or vascular obstruction on the side of planned study access creation, unless corrected prior to randomization
* Planned arteriovenous fistula creation by means other than suture or vascular anastomotic clips (e.g. endovascular surgery or other anastomotic creation devices)
* Anticipated kidney transplant within 12 months
* Anticipated conversion to peritoneal dialysis within 12 months
* Anticipated transfer of nephrology care to a clinic outside the study participating centers within 12 months
* Anticipated non-compliance with medical care based on physician judgment
* A condition in which, in the opinion of the site PI renders the patient not a good candidate for study participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Catheter-free dialysis days | Until death, collected up to 4 years
  Determine the effects of arteriovenous (AV) fistula vs. AV graft vascular access strategy on the rate of catheter-free dialysis days
Number of Infections | Until death, collected up to 4 years
  Access-related infections - catheter-related blood-stream infection, with or without sepsis, requiring hospitalization for treatment

SECONDARY OUTCOMES:
Vascular access-related cost per patient-year | Year 2
  The total cost will represent the sum of costs for adjuvant procedures (endovascular and surgical) related to fistula or graft access; central venous catheter (CVC) - related interventions; infectious complications related to fistula or graft access; infectious complications related to CVC; and hospitalizations related to fistula or graft access and/or CVC. All access-related costs will be expressed as mean cost (in U.S. dollars) per patient per year
Incidence rate of study fistula/graft primary maturation failure | hour 72, Month 3, Month 6, and Year 4
  Study fistula or graft primary maturation failure is defined as permanent failure of the fistula or graft before hemodialysis suitability, and the study fistula or graft access was abandoned. Causes of fistula or graft primary maturation failure include inadequate vasculature, thrombosis, inability to achieve successful cannulation, and other complications leading to nonfunctional fistula or graft - Abandonment of the study fistula or graft access is defined as the point at which the fistula or graft access cannot be cannulated and no further attempts will be made to rescue or revise the access
Time to successful fistula/graft access cannulation | Until death, collected up to 4 years
  This is the time from the date of surgical creation of study AV access (fistula or graft) to the date of successful access cannulation. The date of successful access cannulation is defined as the date when the study fistula or graft access became the primary vascular access for hemodialysis (i.e., the fistula or graft access became the sole vascular access for hemodialysis and the CVC was removed)
Incidence rate of fistula/graft access hemodialysis suitability | Month 6
  Study AV access use (fistula or graft) with two needles for at least 8 out of 12 hemodialysis sessions occurring during the 30-day suitability ascertainment period
Functional patency of study fistula or graft access | Until death, collected up to 4 years
  Total duration of successful use of the study fistula or graft access (i.e., the study fistula or graft access was the sole means of hemodialysis vascular access)
Rate of adjuvant endovascular and surgical procedures | Until death, collected up to 4 years
  All endovascular and surgical procedures performed to evaluate the study fistula or graft access, or to aid or maintain study fistula or graft access functional patency will be included in this outcome. Adjuvant endovascular interventions include: percutaneous thrombectomy; percutaneous revision of anastomosis or dilation of vein/artery (e.g., angioplasty) with or without stent placement; and dilation of central venous stenosis. Adjuvant surgical interventions include: surgical thrombectomy; dilation of central venous stenosis; surgical revision of anastomosis or dilation of vein/artery (e.g., angioplasty) with or without stent placement; ligation of tributaries; superficialization of study fistula; second-stage planned procedure for brachio-basilic fistula creation; ligation of fistula or salvage by distal reconstruction and interval ligation due to distal ischemia.

OTHER OUTCOMES:
Vascular Access Score | baseline and Months 6 and 12
  Satisfaction with different processes of vascular access care (catheter, fistula, or graft) - vascular access questionnaire (VAQ) - satisfaction with the vascular access using the vascular access questionnaire - patient-reported questionnaire composed of 17 vascular access related questions with responses on a five-point Likert scale which are summed, to give a Vascular Access Score- Score range is 4 to 20, with lower scores indicating more satisfaction with the vascular access
SUPPORT Trial questionnaire | baseline and Months 6, and 12
  Will be based on the SUPPORT Trial questionnaire which has two items. The first question asks patients to choose their top priority, extension of life or relieving discomfort as much as possible. The second question asks patients to use the same categories to describe the focus of AV access care they received - This questionnaire will be analyzed using qualitative methods
Decision Regret Scale | Months 6, and 12
  Measuring the regret of AV access placement will be assessed using the Decision Regret Scale - The Decision Regret Scale is a 5-item Likert-type measure written to assess regret or remorse following a medical decision. Patients respond to the items after reading the prompt: "Please think about the decision you made about [chosen health care decision] after talking to your [doctor, surgeon, nurse, health professional, etc.]." High scores suggest high regret over a health care decision. Scores may be transformed to a scale of 0 (no regret) to 100 (high regret)
Attitude Scale | Months 6, and 12
  Participant's preferences between quantity and quality of life and future/present health using the Attitude Scale - An attitude scale is designed to provide a valid, or accurate, measure of an individual's social attitude - The Attitude Scale is composed of 9 items in which participants are asked to rate the strength of the statements, each representing a tradeoff between quality and quantity of life; total score range 9 to 45, with higher scores denoting that quality of life/current health is more important than quantity of life/future health
Grip strength | Months 1, 6, and 12
  Assessed with upper arm grip-strength test in each arm using a hand-held dynamometer - A dynamometer provides objective grip strength data. Males normally can generate about 46 kg of force, and females about 23 kg - A cut-off point <16 kg in women and <26 kg in men will define muscle weakness
Chair stand test | Months 1, 6, and 12
  The chair stand testing will be a timed repetition of rising from a chair and sitting down five times. The test will be scored based on the time (seconds) it takes to complete the five consecutive stand-up-sit-down workouts - longer times denotes worse outcomes. The score ranges from 0 to 4 based on pre-established time cut-offs: 4 points if ≤11.19 sec, 3 points if 11.20-13.69 sec, 2 points if 13.70-16.69 sec, 1 point if ≥16.70 sec, and 0 points if >60 sec or unable.
Clinical Frailty Scale | Months 1, 6, and 12
  Participant's level of frailty using the Clinical Frailty Scale - The Clinical Frailty Scale (CFS) is a judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill) -The scale will be graded from 1 to 7 (1, severely frail; 2, moderately frail; 3, mildly frail; 4, apparently vulnerable; 5, well with treated comorbid disease; 6, well without active disease; 7, very fit
Pepper Assessment Tool for Disability (PAT-D) | Months 1, 6, and 12
  Self-report disability questionnaire using the Pepper Assessment Tool for Disability - The PAT-D self-administered questionnaire consists of 23 items that include a range of activities that assess mobility, activities of daily living (ADL) and instrumental activities of daily living (IADL). For each item, respondents answer whether they experience (1) unable to do, (2) a lot of difficulty, (3) some difficulty, (4) a little difficulty, (5) no difficulty. The summary score, a mean of the three domain scores that ranges from 1 to 5, is an indication of a person's overall perceived disability.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Murea, MD, Principal Investigator — Wake Forest Health Sciences; Matthew P Goldman, MD, Principal Investigator — Wake Forest University Health Sciences; Michael Allon, MD, Principal Investigator — University of Alabama at Birmingham
Locations (7):
- United States (7):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Atrium Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Prisma Health Upstate, Greenville, South Carolina
  - University of Tennessee Medical Center at Knoxville, Knoxville, Tennessee
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Available upon investigator request

REFERENCES:
- [Derived] Murea M, Gardezi AI, Goldman MP, Hicks CW, Lee T, Middleton JP, Shingarev R, Vachharajani TJ, Woo K, Abdelnour LM, Bennett KM, Geetha D, Kirksey L, Southerland KW, Young CJ, Brown WM, Bahnson J, Chen H, Allon M. Study protocol of a randomized controlled trial of fistula vs. graft arteriovenous vascular access in older adults with end-stage kidney disease on hemodialysis: the AV access trial. BMC Nephrol. 2023 Feb 24;24(1):43. doi: 10.1186/s12882-023-03086-5. PMID 36829135